CLINICAL TRIAL: NCT07003113
Title: Ischemic Preconditioning in Osteoarthritis and Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-0021; 90SFE0071 (Other Grant/Funding Number: National Institute on Disability, Independent Living, and Rehabilitation Research)
Record Dates: First submitted 2025-05-23; First posted 2025-06-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain; Knee Osteoarthritis
Keywords: ischemic preconditioning; restricted blood flow; knee pain; back pain
MeSH Terms: conditions — Low Back Pain; Osteoarthritis, Knee; Back Pain | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IC Arm (Experimental)
  Interventions: Device: Ischemic Preconditioning
- Sham Arm (Sham Comparator)
  Interventions: Device: Sham Intervention

INTERVENTIONS:
Device: Ischemic Preconditioning — The intervention arm will include full blood flow occlusion in one thigh for 5 minutes followed by 5 minutes of reperfusion for a cycle of 50 minutes.
  Arms: IC Arm
Device: Sham Intervention — This intervention includes 25mmHg of pressure, which is not sufficient for blodo flow occlusion.
  Arms: Sham Arm

SUMMARY:
We are examining the use of restricted blood flow, through full occlusion, on a single thigh for 50 minutes (5 minutes on, 5 minutes off), completed every other day for 2 weeks to improve function in individuals with knee osteoarthritis and low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Reported Knee Pain using ACR Criteria
* Reported Back Pain using ODI Criteria > 12
* Ability to walk for at least 3 minutes without the use of aids
* Ability to provide written informed consent

Exclusion Criteria:

* Younger than 50 years old
* History of Knee or Hip Replacements
* History of steroid injection within the previous 6 months
* Presence of neuromuscular joint condition that affects lower extremity function
* History of blood clots in the leg or any condition in which compression of the thigh is contraindicated
* History of heart failure or thrombosis
* Allergic to ultrasound gel
* History of spine surgery
* Non-English speaker
* Currently pregnant or intends to become pregnant during the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Preferred walking speed | At baseline (from enrollment) until end of intervention (3 weeks).
  Changes in preferred walking speed (m/s) from intervention
Muscle strength | From baseline (enrollment) until end of intervention (3 weeks)
  Change in quadriceps, hamstring, and hip strength
Patient Reported Outcomes | At baseline (enrollment) through the intervention (3 weeks)
  Change in subjective function and reporting based on questionnaires
Gait Kinematics | At baseline (from enrollment) until end of intervention (3 weeks).
  Changes in gait kinematics (in degrees) from intervention
Gait Kinetics/Moments | At baseline (from enrollment) until end of intervention (3 weeks).
  Changes in gait kinetics (joint moments) (in N/m) from intervention

SECONDARY OUTCOMES:
Cartilage Health | From baseline (enrollment) until completion of intervention (3 weeks)
  Change in knee cartilage thickness using ultrasound methods

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Hannigan, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Human and Sport Performance Lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No